CLINICAL TRIAL: NCT03104101
Title: Evaluation of Transcutaneous Posterior Tibial Nerve Electro Stimulation With or Without Low Dose Trospium Chloride in the Management of Overactive Bladder in Females
Brief Title: Transcutaneous Posterior Tibial Nerve Electrostimulation With Low Dose Trospium Chloride in OAB in Females
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Amr Gaber Abdulfattah Ali Abulseoud, Urology Specialist, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Alexandria University
Record Dates: First submitted 2017-03-09; First posted 2017-04-07 (Actual); Last update posted 2017-04-07 (Actual); Status verified 2017-03

CONDITIONS: Overactive Bladder
Keywords: PTNS; Neuromodulation; TPTNS; Trospium chloride
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TPTNS (Active Comparator): Those who received Transcutaneous posterior tibial nerve stimulation sessions only
  Interventions: Device: TPTNS
- TPTNS+Drug (Active Comparator): Those who received Transcutaneous posterior tibial nerve stimulation sessions plus 20 mg Trospium chloride
  Interventions: Combination Product: TPTNS+Drug

INTERVENTIONS:
Combination Product: TPTNS+Drug — one tablet Trospium Chloride 20 mg once daily Plus TPTNS
  Arms: TPTNS+Drug
Device: TPTNS — Surface adhesive electrodes placed on the skin above medial malleolus
  Arms: TPTNS

SUMMARY:
This study was done to verify whether the combination of transcutaneous posterior tibial nerve stimulation (TPTNS) with low dose trospium chloride in the treatment of females with overactive bladder (OAB) would be more effective than TPTNS alone after failure of behavioral therapy.

DETAILED DESCRIPTION:
The investigators randomized 30 women with OAB, in two groups: G I (15 patients) received 30 minutes TPTNS, three times a week; GII (15 patients) received TPTNS plus Low dose trospium chloride (20 mg once daily); all for 8 weeks. Patients were evaluated using Overactive Bladder Symptom Score questionnaire (OABSS), Incontinence Impact Questionnaire-short form 7 (IIQ-7), 3 day voiding diary and urodynamics at weeks 0 and 8.

ELIGIBILITY:
Inclusion Criteria:

* Thirty adult female patients having OAB symptoms (wet type) and proved to have detrusor overactivity by urodynamics

Exclusion Criteria:

1. Patients having urinary tract infection or bladder outlet obstruction.
2. Patients having neurological diseases.
3. Patients having gynecological problems as genital infection, pelvic organ prolapse or genital tumors.
4. Patients with electronic implants such as heart pacemakers.
5. During pregnancy
6. Patients subject to seizures

Ages: 20 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-11-01 (Actual); Primary Completion 2015-11-30 (Actual); Study Completion 2016-03-05 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction | 1 year
  Improvement in the questionnaire scores and associated willingness of the patient to continue treatment

IPD SHARING:
Plan to Share IPD: Yes